CLINICAL TRIAL: NCT01482897
Title: Open Randomized Study on the Efficacy of corticoïd Infiltration Versus Physiological Solution Infiltration Versus Feigning of Infiltration Via Sacro-coccygien Hiatus Versus Natural Evolution in Discal Sciatica
Brief Title: Efficacy of corticoïd Infiltration Via Sacro-coccygien Hiatus in Discal Sciatica
Acronym: Hiatus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrolment stopped on December 01, 2014 since after 3 years, only 13 patients were included (instead of 274) (Date of last visit last patient : October 3, 2013).
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRD 11/4-M
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Discal Sciatica
Keywords: Discal sciatica, infiltrations; Subjects; evolving
MeSH Terms: interventions — prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- corticoïd (Experimental): anesthetic bloc (10 ml of xylocaïne 1%) immediately followed with corticoid (125mg in.5 ml)
  Interventions: Drug: Prednisolone acetate
- physiological solution (Placebo Comparator): anesthetic bloc (10 ml of xylocaïne 1%) immediately followed with physiological solution (20 ml)
  Interventions: Drug: comparator : physiological solution
- feigning of peridural infiltration (Sham Comparator): feigning of peridural infiltration : anesthetic bloc (10 ml of xylocaïne 1%) immediately followed with placement of empty syringe in peridural.
  Interventions: Drug: sham procedure
- no intervention (No Intervention): natural evolution of discal sciatica

INTERVENTIONS:
Drug: Prednisolone acetate — anesthetic bloc (10 ml of xylocaïne 1%) immediately followed with corticoid (125mg in.5 ml)
  Arms: corticoïd
Drug: sham procedure — feigning of peridural infiltration : anesthetic bloc (10 ml of xylocaïne 1%) immediately followed with placement of empty syringe in peridural.
  Arms: feigning of peridural infiltration
Drug: comparator : physiological solution — anesthetic bloc (10 ml of xylocaïne 1%) immediately followed with physiological solution (20 ml)
  Arms: physiological solution

SUMMARY:
The specific aim of this study is to determine whether a medical intervention improve status of patients with discal sciatica and if yes which type of intervention.

DETAILED DESCRIPTION:
The primary criteria is to determine the difference between the mean leg pain during the latest 24 hours preceding the infiltration and the mean leg pain preceding the visit S4 (visit 4 weeks after the infiltration). If difference is of 50% patient will be considered "improved". This study will be organized under three steps:Step 1 : when 124 patients will be randomized: first intermediate analysis to compare efficacy of groups 1+ 2+ 3 versus 4. If significant difference is not demonstrated, study will be stopped at this stage since having demonstrating that infiltration or simulation is inefficient. On the other case, step 2 will be performed.Step 2 : Recruitment is continued only in arms 1 to 3 until reaching a total of 142 randomized patients. Second intermediate analysis to compare efficacy of groups 1+ 2 versus 3. If significant difference is not demonstrated, study will be stopped at this stage since having demonstrating that infiltration is inefficient. On the other case, step 3 will be performed.Step 3 : Recruitment is continued only in arms 1 and 2 until reaching a total of 274 randomized patients. Third intermediate analysis to compare efficacy of groups 1 versus 2.

Visit of inclusion (J0): 1/ notification in the case report form of - information concerning patient pain (mean, maximal and minimal pain during the 24 last hours)- Oswestry questionnaire - impact of discal sciatica on professional activity,- intake of analgesic, co-analgesics and non steroids anti- inflammatory drugs2/ Randomization and infiltration with corresponding treatment arm3/ Thirty minutes after receiving the infiltration, recording of actual patient pain Visits at day 7, weeks 4, 12 and 24 after J0: Notification in the case report form of - information concerning patient pain (mean, maximal and minimal pain during the 24 last hours)- Oswestry questionnaire - impact of discal sciatica on professional activity,- intake of analgesic, co-analgesics and non steroids anti- inflammatory drugs

ELIGIBILITY:
Inclusion Criteria:

* Adult with age equal or above to 18.
* Subject affiliated to French health insurance (Sécurité Sociale)
* Sciatic pain evolving since more than 1 month and less than 3 months
* Leg irradiation (pain above the knee)- True Lasègue- Mean leg pain during the latest 24 hours above 40 on an analogic visual scale (from 0 to 100)
* Pain induced by palpation in regards to the neo-articulation
* Pain not relieved by medical treatment with non steroids anti- inflammatory drugs or antalgics No sign of seriousness : no motor deficiency (muscular testing above or equal to 4 on an international scale (from 0 to 5), no sphincter deficiency, mean leg pain during the latest 24 hours below 80 on an analogic visual scale (from 0 to 100).
* Scanner of MRI since less than 3 months confirming discal hernia L4L5 or L5S1 in accordance with the clinic.
* Informed consent form signed

Exclusion Criteria:

* Age below 18
* Clinical arguments in favour of a non discal origin- Pregnant women
* Diabetic patient- Past history of diverticulosis complicated with severe arterial hypertension- Patient unable to understand the protocol
* No autonomy for coming to the hospital (no budget allocated for patient transportation)
* Hypersensitivity to local anesthetics with "liaison amide"-Hypersensitivity to one of the components-Porphyria
* Local or generalized infection, suspicion of infection
* Severe troubles of coagulation, anti-coagulant treatment taken- Imaging non concording
* Past history of infiltration via the sacro-coccygien hiatus
* Past history of lombar rachis surgery- Body mass index above 40.
* Intake of "b-bloquants"- Intake of antiarrythmics possibly giving "torsades de pointe" ("amiodarone, disopyramide, quinidiniques, sotalol,…)"-"Cimétidine" used at doses above or equal to 800mg/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
difference between the mean leg pain during the latest 24 hours preceding the infiltration and that preceding the visit S4 | week 4
  To determine the difference between the mean leg pain during the latest 24 hours preceding the infiltration and the mean leg pain preceding the visit S4 (visit 4 weeks after the infiltration). If difference is of 50% patient will be considered "improved".

SECONDARY OUTCOMES:
determine whether medical intervention improve status of patients
  To determine whether:- injection of physiological solution or of physiological solution +hydrocortancyl is more efficient than simple feigning of peridural infiltration
determine whether medical intervention improve status of patients
  to determine wheter the improvement by the infiltration of corticoid is present at visit of 7 days after the infiltration and at visits of 3 and 6 months after the infiltration
To determine whether intervention can decrease the number of surgeries (follow-up of 6 months)
  To determine whether intervention can decrease the number of surgeries (follow-up of 6 months)
To determine whether intervention can decrease the intake of drugs
  to determine whether intervention can decrease the intake of drugs
To determine whether intervention can decrease the functional handicap
  To determine whether intervention can decrease the functional handicap

CONTACTS AND LOCATIONS:
Overall Officials: Joelle Glemarec, Doctor, Principal Investigator — CHU of Nantes; Grégoire CORMIER, Doctor, Principal Investigator — CHD of La Roche/Yon
Locations (1):
- Universitary Hospital, Nantes, Loire Atlantique, France